CLINICAL TRIAL: NCT01551394
Title: Efficacy, Pharmacokinetics and Safety of Meropenem in Infants Below 90 Days of Age (Inclusive) With Clinical or Confirmed Late-onset Sepsis : a European Multicenter Randomised Phase III Trial
Brief Title: Efficacy, Pharmacokinetics and Safety of Meropenem in Infants Below 90 Days With Clinical or Confirmed Late-onset Sepsis
Acronym: NeoMero-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-001515-31
Record Dates: First submitted 2012-02-27; First posted 2012-03-12 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Sepsis
Keywords: sepsis; neonates; meropenem
MeSH Terms: conditions — Sepsis | interventions — Meropenem; Ampicillin; Gentamicins; Cefotaxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meropenem (Experimental): Infants will received the Meropenem 20 mg/kg every 8 hours (every 12 hours in the youngest age group: < 32 weeks GA and < 2 weeks postnatal age). The dose will be given as an infusion over 30 minutes.
  Treatment duration is 11 ± 3 days.
  Interventions: Drug: Meropenem
- Standard of care (Active Comparator): The two accepted therapeutic options are:
  * ampicillin + gentamicin (SOC regimen 1) and
  * cefotaxime + gentamicin (SOC regimen 2).
  Interventions: Drug: Ampicillin + gentamicin or cefotaxime + gentamicin

INTERVENTIONS:
Drug: Meropenem — 20 mg/kg every 8 hours (every 12 hours in the youngest age group: < 32 weeks GA and < 2 weeks postnatal age). The dose will be given as an infusion over 30 minutes. Treatment duration is 11 ± 3 days.
  Other Names: Meropenem trihydrate
  Arms: Meropenem
Drug: Ampicillin + gentamicin or cefotaxime + gentamicin — Ampicillin:
  Neonates below 7 days: 50mg/kg every 12 hours Neonates 7-21 days: 50mg/kg every 8 hours Neonates and Infants from day 22 on: 50mg/kg every 6 hours
  Gentamicin:
  Neonates less than 32 weeks of corrected age: 5mg/kg every 36 hours Neonates 32 weeks and over of corrected age: 5mg/kg every 24 hours (pre-dose ('trough') concentrations should be less than 2mg/l) Infants over 28 days of postnatal age: once daily dose: initially 5-7mg/kg, then adjust according to serum-gentamicin concentration (pre-dose ('trough') concentrations should be less than 1mg/l)
  Cefotaxime:
  Neonates below 7 days of PNA: 50mg/kg every 12 hours Neonates and infants from day 7 of PNA: 50mg/kg every 8 hours Treatment duration is 11 ± 3 days.
  Other Names: Ampicillin sodium; Gentamicin sulphate; Cefotaxime sodium
  Arms: Standard of care

SUMMARY:
This phase III multicentric international randomized trial is designed to compare the efficacy of Meropenem to the standard of care in infants below 90 days of age with clinical or confirmed late-onset sepsis (LOS).

The aim is to assess efficacy , pharmacokinetics and safety of Meropenem which are not well known and documented in this population.

DETAILED DESCRIPTION:
The principal objective is to compare the efficacy at test of cure (TOC) visit of meropenem to the standard of care (SOC) in the treatment of clinical or confirmed LOS in infants ≤ 90 days of postnatal age.

The secondary objectives are:

* To compare the safety profile of meropenem to SOC
* To compare the efficacy at TOC visit of meropenem to SOC in confirmed sepsis
* To compare the response to meropenem and SOC on day 3 of antibacterial therapy
* To compare the efficacy at TOC visit of meropenem to SOC ignoring the change of antibiotic(s) for safety reasons
* To compare the efficacy at TOC visit of meropenem to SOC by SOC regimen
* To compare survival at follow up (FU) visit (28 day visit) in the meropenem arm and SOC arm
* To compare new infections and relapses that occur between TOC and FU visits in participants with a favourable outcome at TOC visit by treatment arm
* To define the organisms causing LOS
* To study antibacterial susceptibility of LOS-causing organisms and to describe clinical and microbiological responses according to this
* To compare gut colonization by antibiotic resistant organisms after treatment with meropenem or SOC
* To compare bacterial eradication by treatment arm
* To compare time to NICU discharge across the 2 arms
* To describe PK of meropenem in infants ≤ 90 days of postnatal age with LOS
* To evaluate genetic parameters that may affect response to therapy

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the parents/carers
* Chronological age below 90 days inclusive
* Chronological age greater or equal to 72 hours of life at beginning of LOS
* Clinical or confirmed sepsis

  * For infants below 44 weeks inclusive of corrected age

clinical sepsis is defined, according to the Expert Meeting on Neonatal and Paediatric Sepsis (Report on the Expert Meeting on Neonatal and Paediatric Sepsis - 8 June 2010, EMA London), as the presence in the last 24 hours of at least

* two clinical criteria:

  * hyper- or hypothermia or temperature instability,
  * reduced urinary output or hypotension or mottled skin or impaired peripheral perfusion
  * apnea or increased oxygen requirement or increased requirement for ventilatory support,
  * bradycardia spells or tachycardia or rhythm instability,
  * feeding intolerance or abdominal distension,
  * lethargy or hypotonia or irritability,
  * skin and subcutaneous lesions such as petechial rash or sclerema,
* and two laboratory criteria:

  * white blood cells (WBC) count < 4 or > 20 x 109 cells/L,
  * immature to total neutrophil ratio (I/T) > 0.2,
  * platelet count < 100 x 109/L,
  * C-reactive protein (CRP) > 15 mg/L or procalcitonin ≥ 2 ng/mL,
  * glucose intolerance when receiving normal glucose amounts (8-15 g/kg/day) as expressed by blood glucose values > 180 mg/dL or hypoglycemia (< 40 mg/dL) confirmed at least two times,
  * acidosis as characterized by base excess (BE) < -10 mmol/L or lactate with value above 2 mmol/L.

confirmed sepsis is defined as positive culture for pathogens in a sample from a normally sterile site and at least one laboratory sign or clinical sign (from the list above)

* For children above 44 weeks corrected age

clinical sepsis is defined according to the Goldstein criteria (Goldstein et al, 2005) as at least two of the following criteria, one of which must be abnormal temperature or WBC count:

* Core temperature of > 38.5 °C or < 36 °C;
* Tachycardia, defined as mean heart rate > to the 95th percentile for age group in the absence of external stimulus, chronic drugs, or painful stimuli or unexplained persistent elevation over a 0.5 to 4 hour time period; or bradycardia, defined as a mean heart rate < to the 5th percentile for age group in the absence of external vagal stimulus, beta blocker drugs, or congenital heart disease or unexplained persistent depression over a 0.5 hour time period;
* Mean respiratory rate > to the 95th percentile for age group or mechanical ventilation for an acute process not related to underlying neuromuscular disease or the receipt of general anaesthesia;
* Leukocyte count < the 5th percentile or > than the 95th percentile for age group (not secondary to chemotherapy-induced leucopoenia).

confirmed sepsis: positive culture for pathogens in a sample from a normally sterile site and at least one laboratory sign or clinical sign (from the list above)

Exclusion Criteria:

* Administration of any systemic antibiotics for more than 24 hours prior to the randomisation, unless the change is driven by the lack of efficacy of the former regimen;
* Severe congenital malformations if the infant is not expected to survive for more than 3 months;
* Other situations where the treating physician considers a different antibiotic regimen necessary;
* Known intolerance or contraindication to study medication;
* Participation in any other clinical study of investigational drugs;
* Renal failure (as defined by Akcan-Arikan et al., 2007) and requirement of haemofiltration or peritoneal dialysis;
* Confirmed sepsis with microorganisms known to be resistant to study therapies.

Ages: 72 Hours to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 272 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
percentage of patients with a favorable outcome in the two arms | an expected average of 14 days
  The proportions of participants with a favourable outcome will be calculated in the meropenem arm and in the SOC arm. A favourable outcome is met when an infant:
  * Is alive
  * Has resolution or significant improvement of all abnormalities that defined LOS at entry and has no new clinical or laboratory abnormalities requiring a new course of antibiotic therapy
  * Has microbiological eradication either confirmed or presumed and no new pathogens identified.

SECONDARY OUTCOMES:
Nature, frequency and numbers of clinical and biological adverse events | 3 - 28 days
  Adverse events will also be summarised according to the need of a specific medical intervention or not. Analyses by time period will also be shown (from D0 to TOC visit and from TOC visit to follow-up). The number of patients experiencing at least one adverse event between D0 and TOC visit will be compared by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Trafojer, Principal Investigator — Clinica Pediatrica, Padova; Irja Lutsar, Principal Investigator — University of Tartu, Estonia; Jean-Pierre Aboulker, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Ursula TRAFOJER, Padua, Italy

REFERENCES:
- See also: Site dedicated to the NeoMero studies — http://www.neomero.org